CLINICAL TRIAL: NCT01248689
Title: The Effect of Different Concentrations of Sevoflorane on Intraocular Pressure in Children Undergoing Ocular Surgery Under General Anesthesia
Brief Title: Effect of Sevoflurane Concentration on Intraocular Pressure in Surgical Children With Healthy Eyes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Professor Idit Matot. Chair, Department of Anesthsiology & Intensive Care, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: TASMC-10-IM-0553-CTIL
Record Dates: First submitted 2010-11-17; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-11

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- concentration profile 1 (Active Comparator): IOP will be measured under this order of sevoflurane concentrations:
  7%, 5%, 2%, 0.5%
  Interventions: Other: concentration profile 1
- concentration profile 2 (Active Comparator): IOP will be measured under this order of sevoflurane concentrations:
  7%, 2%, 5%, 0.5%
  Interventions: Other: concentration profile 2
- concentration profile 3 (Active Comparator): IOP will be measured under this order of sevoflurane concentrations:
  7%, 0.5%, 5%, 2%
  Interventions: Other: concentration profile 3

INTERVENTIONS:
Other: concentration profile 1 — IOP will be measured under this order of sevoflurane concentrations:
  7%, 5%, 2%, 0.5%
  Other Names: IOP measurements 1
  Arms: concentration profile 1
Other: concentration profile 2 — IOP will be measured under this order of sevoflurane concentrations:
  7%, 2%, 5%, 0.5%
  Other Names: IOP measurements 2
  Arms: concentration profile 2
Other: concentration profile 3 — IOP will be measured under this order of sevoflurane concentrations:
  7%, 0.5%, 5%, 2%
  Other Names: IOP measurements 3
  Arms: concentration profile 3

SUMMARY:
One important goal in anesthetic management during ocular surgery is to provide adequate control of intraocular pressure (IOP). An increase in IOP may be catastrophic in patients with glaucoma or a penetrating open-eye injury. Accurate assessment of IOP is particularly important in infants and children with definite or suspected glaucoma undergoing examination under anesthesia.

Anesthetic regimens in this surgical field commonly consist of short-acting anesthetic agents, such as sevoflurane. Sevoflurane is known to reduce the IOP. During pediatric ocular surgery, the inspired sevoflurane concentration varies continuously and may have an impact over the IOP that could affect the conduct of surgery. In this study the investigators wish to evaluate whether variations in sevoflurane concentration do affect the IOP.

DETAILED DESCRIPTION:
Introduction One important goal in anesthetic management during ocular surgery is to provide adequate control of intraocular pressure (IOP). An increase in IOP may be catastrophic in patients with glaucoma or a penetrating open-eye injury. Accurate assessment of IOP is particularly important in infants and children with definite or suspected glaucoma undergoing examination under anesthesia (EUA).

There is an ongoing debate over the effect of anesthetic agents on the IOP. Anesthetic regimens in this surgical field commonly consist of short-acting anesthetic agents, such as propofol and sevoflurane, usually combined with short-acting analgesics, such as remifentanil [1-3].

Both propofol and sevoflurane are known to reduce the IOP [4-7]. Previous studies have compared these two anesthetics protocols in order to determine which provides superior control of the IOP. Propofol produced significantly lower IOP measurements compared to sevoflurane (both combined with remifentanil), in cataract surgery [8], whereas in non-ophthalmic surgery propofol and sevoflurane caused a comparable decrease in IOP [9].

Sevoflurane, an inhalational anesthetic, has a rapid onset of action, faster recovery time and lower incidence of reported side effects in pediatric patients [10], and is also suitable for inhalation induction because it does not irritate the airway [3].

During pediatric ocular surgery, the inspired sevoflurane concentration is normally maximal at induction of anesthesia (approximately end-tidal concentration of 7%), and it is thereafter reduced or discontinued to achieve an end-tidal sevoflurane concentration of <0.1% by the completion of skin closure. In between these time points the inhaled end-tidal concentration gradually decreases and may have an impact over the IOP that could affect the conduct of surgery. A prospective randomized clinical trial compared the effects of ketamine and sevoflurane on IOP during the eight minutes after induction of anesthesia (in 2-minute intervals) in children with suspected or diagnosed glaucoma undergoing EUA [5]. During these 8 minutes the IOP decreased significantly only in the sevoflurane group. This finding contradicted claims that measurements immediately after induction are relatively unaffected by anesthetics, and suggested that variations in sevoflurane concentration do affect the IOP. To this end there is no data in the literature to support or disprove this finding.

Study Objective To assess the effect of different end-tidal sevoflurane concentrations on the IOP in children with healthy eyes undergoing extraocular procedures, i.e., strabismus correction and tear duct probing and irrigation.

Study hypothesis We believe that variations in the end-tidal sevoflurane concentrations have no significant effect on the IOP of healthy eyes.

Study design This is a prospective randomized trial of 21 children undergoing ocular surgery. Informed consent will first be obtained from the parent or legal guardian. After induction of anesthesia and before onset of surgery, IOP will be measured in both eyes under four different concentrations of inhaled sevoflurane.

Intra-operative anesthetic management Anesthetic management will be performed by a trained pediatric anesthesiologist. All patients will be premedicated with 0.5 mg/kg (up to 15 mg) midazolam P.O. 30min before surgery. No significant change in IOP has been reported for midazolam [11]. Induction of anesthesia will be carried out with sevoflurane 8% in 100% oxygen carrier gas. After induction of anesthesia, laryngeal mask will be inserted, and sevoflurane end-tidal concentrations will be adjusted according to the study protocol and assigned group (see "patient allocation and assessment"). No other systemic anesthetic agents will be used during IOP measurements. IOP measurements will be performed after induction of anesthesia. Thereafter, maintenance of anesthesia will be carried out with either spontaneous ventilation at one to two minimal alveolar concentration of sevoflurane (2 to 4%) in 100% oxygen, or mechanical ventilation, as commonly used in pediatric surgery. Standardized intraoperative monitoring will be employed for all subjects by an anesthesiologist.

Intra-operative surgical management Routine strabismus correction or tear duct probing and irrigation procedures will be performed on each subject, as described elsewhere [12].

Patient allocation and assessment

Consented patients will be randomly (by means of computer-generated assignment of random numbers) allocated to one of three groups (n=7 in each group). In each group IOP will be measured and recorded under four different predetermined end-tidal sevoflurane concentrations: 7%, 5%, 2%, 0.5%. The order of concentrations will differ between the groups, to eliminate the effect of exposure time:

1. 7%, 5%, 2%, 0.5%
2. 7%, 2%, 5%, 0.5%
3. 7%, 0.5%, 5%, 2% IOP will be measured by the ophthalmologist via both TonoPen XL and Schioz devices. Measurements will be taken from each eye alternatively for three consecutive readings, at each of the abovementioned concentrations. There is no known risk at IOP reading. At the same times, the anesthesiologist will record systolic and diastolic blood pressure (SBP, DBP) and heart rate (HR), End Tidal CO2, via iMDsoft software.

In addition, we will collect demographic data (e.g., age, gender, weight) for each patient. Routine post operative follow up will be performed.

ELIGIBILITY:
Inclusion Criteria:

* children with healthy eyes, undergoing elective surgery for strabismus correction or tear duct probing and irrigation.

Exclusion Criteria:

* children with adverse reaction or contraindication (of any other reason) to sevoflurane or remifentanil, and patients with pre-existing intra-ocular ophthalmic disease, or infection.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
IOP | first hour of anesthesia
  IOP will be measured in both eyes, after induction of anesthesia and before the onset of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, MD, Study Chair — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Artru AA, Momota Y. Trabecular outflow facility and formation rate of aqueous humor during anesthesia with sevoflurane-nitrous oxide or sevoflurane-remifentanil in rabbits. Anesth Analg. 1999 Apr;88(4):781-6. doi: 10.1097/00000539-199904000-00019. PMID 10195524